CLINICAL TRIAL: NCT02002520
Title: An Exploratory Study of the Epigenetic Influences on Post-Surgical Acute and Chronic Pain
Brief Title: Epigenetic Influences on Post-Surgical Acute and Chronic Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheung Chi Wai, Associate Professor, The University of Hong Kong
Other Study IDs: UW13-354
Record Dates: First submitted 2013-11-30; First posted 2013-12-06 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Acute Pain
Keywords: Acute pain; Epigenetic; Dental pain
MeSH Terms: conditions — Acute Pain; Toothache

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — RNA and DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- case group: patients undergo third molar surgery
- control group: subjects do not require surgery

SUMMARY:
Pain is the way our brain interprets certain bodily sensations. It is very difficult to describe or to put into words as perception and tolerance of pain varies widely between individuals. It is known that age, gender and past experience and memory of past experience all contribute to patients' feelings of discomfort and tolerance of pain, but the reason why some patients actually do not experience any pain at all post surgery is still unknown.

Because pain affects every person at some point in their lives, it is of utmost importance that we can find more effective analgesic methods, and provide analgesia tailored to an individual's need as well as discovering new methods which may be able to identify those individuals who are more prone to suffering serious, or chronic pain. It has been proposed that epigenetic modifications may play a role in sensitivity to analgesia and response to trauma, such as post surgery. The effects of epigenetic changes on key genes and the role this plays in analgesia sensitivity and pain perception is deserving of further research.

Epigenetics is a growing field of study in which there are genetic modifications that do not involve changes to base sequences in a gene, but that result nonetheless in changes to gene expression. It has long been known that changes in gene expression play an important role in the establishment of pain states. But it is not known whether a priming injury can induce lasting epigenetic marks which would result in an increase in both postoperative acute pain and the risk for chronic pain. Only by fully understanding these epigenetic mechanisms will we be able to offer better drugs for the treatment of pain, and to identify those at high risk of postoperative pain and postsurgical chronic pain.

The purpose of this study is to determine whether severity of pain following surgical procedures, such as third molar surgery is related to baseline methylation status of the promoter region of IL-6 and TNF-α and changes in methylation status post surgery.

DETAILED DESCRIPTION:
(i) Subjects: Sixty subjects who will be undergoing third molar surgery (hereafter known as 'cases') will be recruited from The Queen Mary Hospital and The Prince Philip Dental Hospital and sixty, aged and sex matched controls who will not be undergoing surgery in the next 3 months, nor have undergone surgery in the past year (hereafter known as 'controls') will also be recruited from the Outpatients department of the same hospital.

(ii) Methods: The study aims and details will be explained to each subject and informed consent will be sought from each of them. A pain diaryquestionnaire developed by our group will be adapted for the use of assessing pain experienced by each subject pre and post surgery. Research personnel will accompany each case subject, and fill out the pain diaryquestionnaire with them during the visit when the patients' blood is taken.

The following health questionaires will be completed by the subjects recruites:

SF-36: 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures HADS: Assessment of the psychological status of the subjects (anxiety & depression)

Pain assessment:

Pain at rest and during opening will be assessed using a numerical rating scale (NRS, 1= no pain, 10 = most severe pain) at the following time points:

1. Before surgery
2. 4 hourly after surgery for 16 hours
3. At 24th, 48th and 72nd after surgery
4. 1 month after surgery by telephone interview.
5. 3 month after surgery by telephone interview. If pain is present, questions about neuropathic pain will be asked.

Venous EDTA blood (10ml) on each occacasion will be drawn from each case one hour prior to surgery, 1 hour and 3 hours post surgery. Then they will be asked to return to the hospital 3 to 5 days post surgery for one more blood taking, and macrophages will be separated from the blood and total RNA will be extracted as soon as possible after blood taking from half the total cells. The remainder of the cells (macrophages) will be stored at -80oC and batched for DNA extraction. Venous EDTA blood (20ml) will be drawn from each control subject at a time convenient to them and again, 3 to 5 days post first blood taking. The blood taken from the control subjects will be treated in exactly the same way as with blood taken from the case subjects. Therefore, four samples in total will be obtained from each case and control subject.

The size of the IL-6 and TNF-α promoter regions spanning the sequences upstream of the transcriptional start site as well as part of the first exon will be determined from literature search and using a database for reference, CpG islands will be first identified for primer design (http://www.cpgislands.com/). For analysis of methylation, a commercial kit will be used (EpiTect Plus LyseAll Bisulfite Kit from Qiagen, Hilden, Germany).

Samples will undergo bisulfite-conversion, and unmethylated cytosines will be deaminated, forming uracils. Methylated cytosines will remain unchanged. The location of the methylated cytosine of the gene sequence and the amount of methylated cytosine will be identified and quantitated by Pyrosequencing using established techniques. Results will be expressed as % methylation in the promoter region of IL-6 and NF-ĸB.

Note: The pyrosequencing technique can only analyse fragments of DNA of up to 50 base pairs in one reaction. According to data from CpG Island Searcher, and when the % GC was set at 55%, observed CpG/expected CpG set at 0.65 and gaps between adjacent islands set at 100bp, no CpG islands can by found in either the IL-6, or the TNFα promoter. Therefore, the methylation status of the whole promoter region in both genes will be studied using 40 pairs of primers for each gene (in order to cover 2kb of the promoter region). This approach is adopted as it is the most sensitive and reliable for determination of site specific DNA methylation in an extended region such as a promoter region.

(iii) Study design: This is a case-control study. The samples used in this study will be whole blood samples taken pre- and post- surgery from the cases, and at a matched time, from the controls.

Power calculations: No data exist on the level of DNA methylation in the promoter region of IL-6 and TNF-α in normal healthy subjects. Power calculations reveal that 51 subjects in each group are required to have an 80% power to detect a true difference in the variable of interest at 5% significance level (calculations using G*Power software, version 3.1). A total of 60 subjects will be recruited into each group to take into consideration drop out rates.

(iv) Data processing and analysis: Paired t-test (or non-parametric equivalent) will be performed to investigate differences in level of DNA methylation pre- and post- surgery. Unpaired t-test will be used to investigate difference in the level of DNA methylation between cases and controls. Correlational analysis will be used to investigate relationships between methylation status and IL-6 and TNF-α expression. Descriptive statistics will be employed to describe the changes in methylation status (i.e., if different sites in the CpG island are methylated) in the promoter region of IL-6 and TNF-α B, pre-post surgery and in the two different sampling time points of the control subjects.

Purpose and potential: This is a pilot, exploratory environmental-epigenetics study on the effect of bilateral third molar surgery on DNA methylation changes in the promoter region of IL-6 and NF-ĸB, and the influence of methylation status on gene expression. The results will provide insight and promote understanding into the molecular mechanisms through which the methylation status of inflammatory genes can affect the experience of pain post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient requires third molar surgery for case group and patient does not require surgery for control group
* Age 18 or above
* Ability to read and understand the study information and consent form
* Written consent obtained

Exclusion Criteria:

* Patient does not requires third molar surgery for case group and patient requires third molar surgery for control group
* Age below 18
* Major cognitive or psychiatric disorders that affect the ability to complete study
* Refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects at Prince Philip Dental Hospital and Queen Mary Hospital
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-09 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
pain score | From postoperative 1 hour to postoperative 3 months

SECONDARY OUTCOMES:
IL-6 and TNF-α expression | From postoperative 1 hr to postoperative 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Chi W Cheung, Principal Investigator — Department of Anaesthesiology, The University of Hong Kong
Locations (1):
- Department of Anaesthesiology, The University of Hong Kong, Hong Kong, Hong Kong